CLINICAL TRIAL: NCT00632268
Title: Phase II Study of Low-dose RAD001(Everolimus) Plus Cisplatin and HDFL (Weekly 24-Hour Infusion of High-dose 5-Fluorouracil and Leucovorin) Chemotherapy for First-line Treatment of Unresectable, Recurrent or Metastatic Gastric Cancer
Brief Title: Low-dose RAD001(Everolimus) Plus Cisplatin-HDFL Chemotherapy for the First-line Treatment of Advanced Gastric Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Collaborators: National Cheng-Kung University Hospital (Other); Taipei Veterans General Hospital, Taiwan (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 200612015M
Record Dates: First submitted 2008-03-03; First posted 2008-03-10 (Estimated); Last update posted 2013-08-21 (Estimated); Status verified 2013-08

CONDITIONS: Metastatic Gastric Cancer
Keywords: mTOR inhibitor; RAD001; everolimus; chemotherapy; cisplatin; high-dose 5-FU
MeSH Terms: conditions — Stomach Neoplasms | interventions — Everolimus; Cisplatin; Fluorouracil; Leucovorin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- A (Experimental): Drug:RAD001 Drug:Cisplatin Drug:5-FU
  Interventions: Drug: RAD001; Cisplatin; 5-FU; Leucovorin

INTERVENTIONS:
Drug: RAD001; Cisplatin; 5-FU; Leucovorin — RAD001: oral 10mg/day on Day 1,8,15 Cisplatin:infusion 35mg/m2/day on Day 1,8 5-FU:infusion 2000mg/m2/day on Day 1,8,15

SUMMARY:
The primary end-point of this study is to evaluate the objective response rates, and the secondary end-points are overall survival, progression-free survival and safety profile of low-dose RAD001 (everolimus) plus cisplatin and HDFL (weekly 24-hour infusion of high-dose 5-FU and leucovorin) chemotherapy in the first-line treatment for patients with unresectable, recurrent, or metastatic gastric cancer.

DETAILED DESCRIPTION:
Non-resectable gastric cancer is an incurable disease, with a median survival of 4 months if untreated. Systemic chemotherapy confers prolongation of survival and improvement of quality of life. Regimens containing cisplatin and 5-fluorouracil (5-FU) are widely adopted in the world. The overall response rate and median overall survival of the P-HDFL regimen (cisplatin and weekly 24-hour infusion of high-dose 5-FU and leucovorin) for advanced gastric cancer are 60% (45%-76%, 95% C.I.) and 10 months, respectively. This regimen (P-HDFL) is very popular in Taiwan because of high objective response rates and low treatment-related toxicities. Adding a third active chemotherapeutic agent to cisplatin and 5-FU doublet does not seem to improve efficacy. Further, most of the patients with recurrent or metastatic gastric cancer are frequently associated with a poor general condition which prohibits intensive chemotherapy. Therefore, combination of P-HDFL with biologic agents(such as everolimus, etc.)is an attractive alternative.

PI3K/Akt/mTOR pathway is actively participating in cell proliferation and survival of human gastric cancers. We have recently demonstrated that RAD001(everolimus),an mTOR inhibitor, although with only modest growth inhibitory effects as a single agent, has significant synergistic cytotoxicity with cisplatin and 5-FU in gastric cancer cells. The concentration of RAD001 needed for synergism with cisplatin and 5-FU is as low as 0.5 to 5 nM. And, as expected, RAD001 has significant inhibition of downstream molecules such as 4E-BP1 and S6Kinase, in human gastric cancer cells. It is therefore reasonable to conduct a phase II study to examine if the combination of a relatively low dose of RAD001 and P-HDFL may improve the outcome of advanced gastric cancer.

This is an open-label, multi-center, phase II trial using low-dose RAD001 (10 mg po on D1,D8,&D15) plus P-HDFL chemotherapy (cisplatin 35 mg/m2 ivd 24 hrs on D1 & D8; 5-FU 2,000 mg/m2 and leucovorin 300 mg/m2 ivd 24 hrs on D1,D8,&D15) in chemotherapy-naïve patients with unresectable locally advanced, recurrent or metastatic gastric cancer. The treatment will be repeated every 28 days. The primary end-point is objective response rates evaluated by RECIST criteria, and the secondary end-points are overall survival, progression-free survival and safety profile. Approximately 41 patients will be enrolled in order to obtain the 37 evaluable patients required by Simon two-stage minimax design. All enrolled patients will be subjected to toxicity evaluations, but optionally to the correlative translational study of biomarkers in peripheral blood mononuclear cells. Patients with massive malignant ascites will optionally participate the study of biomarkers in neoplastic cells in ascites.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have a histologically proven adenocarcinoma of the stomach, with unresectable locally advanced, recurrent or metastatic disease;
2. Patients must receive no prior chemotherapy for unresectable locally advanced, recurrent or metastatic gastric cancer. Previous post-gastrectomy adjuvant therapy should be completed more than 6 months before enrollment;
3. Patients must have at least one "measurable" lesion (by RECIST);
4. Patients must have adequate baseline organ functions, and fasting triglyceride level >/= 70 mg/mL;
5. Patients must be younger than 75 years of age;
6. Patients must have an ECOG performance status </= 2;
7. Patients' life expectancy should be expected >/= 3 months;
8. Patients must sign an informed consent form.

Exclusion Criteria:

1. Patients who have received radiotherapy, chemotherapy, or other experimental therapy within the previous 4 weeks or who are planning to receive such therapies simultaneously with RAD001 plus P-HDFL;
2. Patients who have known hypersensitivity to everolimus, sirolimus or to its derivative;
3. Patients who should not withdrawal from medication which can induce or inhibit activity of CYP3A4 during study period;
4. Patients who have uncontrolled concurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations;
5. Patients with CNS metastasis;
6. Patients who refuse port-A implantation;
7. Women who are currently pregnant or breast feeding, and women of child-bearing potential without adequate contraception;
8. Patients who have another prior malignancy, except for adequately treated basal cell, cervical carcinoma in situ, or any cancer from which the patient has been disease-free for 5 years.

Max Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2008-02; Primary Completion 2012-09 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
To evaluate the confirmed objective response rates (complete and partial responses) | 2008 ~2009

SECONDARY OUTCOMES:
To assess the overall survival(OS), progression-free survival(PFS), treatment-related toxicities, and pharmacokinetic profile of RAD001 used in combination with 5-FU and cisplatin | 2009~2010

CONTACTS AND LOCATIONS:
Overall Officials: Kun-Huei Yeh, M.D.,Ph.D., Principal Investigator — Department of Oncology, National Taiwan University Hospital
Locations (1):
- Department of Oncology, National Taiwan University Hospital, Taipei, Taiwan